CLINICAL TRIAL: NCT06817759
Title: Study Protocol for the Development of an Intervention Integrating Procedures Combining Hypnosis and Virtual Reality in the Support of Patients with Myeloma and Lymphoma During Stem Cell Transplant: a Pilot Randomized Clinical Trial
Brief Title: Development of an Intervention Integrating Procedures Combining Hypnosis and Virtual Reality in the Support of Patients with Hematological Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-3251
Record Dates: First submitted 2025-01-27; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Blood Cancer; Multiple Myeloma (MM); Lymphoma
Keywords: Virtual reality hypnosis; Quality of life; Blood cancer; Oncology; multiple myeloma; lymphoma; hypnosis; virtual reality; hematology; anxiety; pain; stem cells transplantation
MeSH Terms: conditions — Hematologic Neoplasms; Multiple Myeloma; Lymphoma; Neoplasms; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: participants will be recruited and randomly assigned to two conditions: VRH, and a control condition (C) (waiting-list, will receive the intervention after the end of the study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (VRH) group (Experimental): Four obligatory accompanied session of VRH and use of VRH as needed.
  Interventions: Device: Virtual Reality Hypnosis; Device: VRH : Beach; Device: VRH : Forest; Device: VRH : MagicHand; Device: VRH : SecurityProtection
- Control group (No Intervention): Standard of care (waiting list, will receive VRH following the study).

INTERVENTIONS:
Device: Virtual Reality Hypnosis — An intervention program (VRH) that combines VR and hypnosis; Can use it whenever and how much they want. It contains 200 landscapes in VR and 4 different VRH sessions
  Arms: Intervention (VRH) group
Device: VRH : Beach — Hypnosis session with a VR immersion at the beach; one accompanied session
  Arms: Intervention (VRH) group
Device: VRH : Forest — Hypnosis session with a VR immersion in forests; one accompanied session
  Arms: Intervention (VRH) group
Device: VRH : MagicHand — Hypnosis session with a VR immersion with techniques to reduce pain; one accompanied session
  Arms: Intervention (VRH) group
Device: VRH : SecurityProtection — Hypnosis session with a VR immersion with techniques to reduce anxiety; one accompanied session
  Arms: Intervention (VRH) group

SUMMARY:
Research into cancer patients has shown that quality of life is significantly altered by the disease and its associated treatments and is also reported to be a predictor of significant emotional distress. Blood cancer patients are among those most affected in terms of quality of life, facing stem cell transplantation after high-dose chemotherapy, a treatment that is recognized as one of the most stressful of cancer therapy, due to the many adverse effects, including pain, and the uncertainty linked to the fear of graft failure. Hypnosis interventions are proving effective in treating common side effects: nausea, pain, fatigue, anxiety, depressive symptoms and improving overall quality of life, and other interventions, based on virtual reality, have shown promising effects on patients' distress and acute pain. The aim of this study is to evaluate the effects of an intervention program combining hypnosis and virtual reality in assisting myeloma and lymphoma patients during stem cell transplantation, with a view to improving their quality of life during this period. The project aims to assess the validity of the intervention, and to evaluate the effects of the intervention on patients' anxiety, pain and fatigue during transplantation. The validity of the intervention will be measured by a questionnaire assessing the relevance and acceptability of the intervention, expected effects, and practical implementation. Socio-demographic and clinical data will be collected from patients, including axiety, pain, fatigue and quality of life, studied at pre (one week after transplantation) and post (one month after transplantation) intervnention, and at follow-up (three month after transplantation).

DETAILED DESCRIPTION:
This proposal aims to reduce anxiety, pain and fatigue of transplant patients and thus improve their quality of life after the end of the intervention. To do this, the investigators will build on studies of VR use in oncology, and thus address the limitations of existing virtual reality (VR) programs, by developing an intervention that combines immersive technologies derived from VR with medical hypnosis (VRH). This new VRH program involves individualized patient management using hypnosis techniques, to promote better absorption into the experience and optimal response to hypnotic suggestions for managing emotions and pain. In concrete terms, this proposal has two complementary objectives:

1. Evaluate the effects of an VRH prototype in reducing anxiety, pain and fatigue in transplant patients, and thus improving their quality of life after the intervention.
2. Gather user experience, satisfaction levels and recommendations for improvement of the VRH prototype from patients

Methods

Intervention: An intervention program (VRH) that combines VR and hypnosis to facilitate the patient's absorption into a safe, benevolent imaginary world, in which they will be invited to live an experience that distracts them from their negative emotions and pain (Toujours Dimanche application).

The virtual experience will be structured along the lines of a hypnosis session: 1- A soothing immersion will first be offered to catalyze absorption through gentle descents and calming audio-visual stimuli, 2- Reaching a safe, relaxing space, dreamily representing two soothing natural environments (beach or park of the patient's choice), 3- Two therapeutic stress-management activities (dropping into a bag containing all the stress the participants want to get rid of, and allowing the participants to be carried by an imaginary horse, which enables them to escape to a safe place), 4- a physical discomfort manipulation activity enabling participants to remove the sensation of discomfort from the part of their body afflicted by it, and 5- Return to an awake state of consciousness.

The application allows the patient to visit a pleasant place either by taking control of it or in a guided way accompanied by a hypnosis verbatim. The patient can choose between these two options, and the investigators document how he or she uses the application.

Participants : Sixty participants with hematological cancer undergoing stem transplantation will be included in this research. They will be randomized in the two groups of the study : VRH and control (waiting list, will have the intervention at the end of the study).

Procedures: Participants will be asked to complete self-evaluations at four measurement points: T0=pre intervention (one week after the day of transplantation), T1=first session (one week after the day of transplantation), T2= one month post-transplantation and T3=three months follow-up post-transplantation. Interviews to gather patient expectations and satisfaction levels will also be conducted at T0 and T3 respectively for patients in the VRH condition. The first session takes place after the transplant (about 1 week) and patients then use the application at their own pace. The headset then remains available for use during the following two weeks. With the application, they have access to 4 hypnosis recordings (Beach, Forest, MagicHand and SecurityProtection) as well as a bank of landscapes they can visit. They have the choice of using contemplative VRH (with hypnosis) or active VR (wandering through the landscapes on their own). How they use the application will be documented with a logbook.

Measures :

Quality of life will be documented by the FACT-BMT, a scale validated for patients undergoing bone marrow transplantation. It contains 50 items divided in 5 subscales : Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, Bone Marrow Transplantation Subscale scored on a 5-points Likert scale.

The HADS, a scale validated in French for cancer, will assess participants' anxiety-depression. This scale is made up of 14 items: 7 items determine the degree of anxiety and the other 7, the degree of depression. The score of each subscale is calculated by summing the score of each item, which varies between 0 and 3, so that each subscale can reach a maximum score of 21

Pain will be assessed with the Brief Pain Inventory. This scale is made of 8 items on a 10-points Lickert scale assessing severity of pain, impact of pain on daily function, location of pain, pain medications and amount of pain relief in the past 24 hours or the past week.

Fatigue will be assessed with the Multidimensional Fatigue Inventory 10 items version (MFI-10) adapted for cancer. It is scored on a 5-points Likert Scale going form 1: "do not agree at all" to 5: "totally agree".

Ten-level Visual Numerical Scales (VNS) will also be used to assess pain, anxiety, absorption, i.e., the tendency to become totally involved in a perceptual and imaginative experience, and dissociation, i.e., a mental separation of components of the experience, fatigue and amusement.

The investigators will collect patients' levels of expectation and satisfaction through 5-level VNS (1 = "not at all satisfied", 5 = "very satisfied") and through explanatory interviews.

The Simulator Sickness Questionnaire, a scale validated in French assesses cybersickness symptoms related to VR immersion. It contains 16 items divided in two subsacles: nausea and oculomotor, which the participant must qualify with "not at all" (scored 0) , "a little" (scored 1), "moderately" (scored 2) or "severely" (scored 3).

Analyses : Continuous quantitative variables will be expressed as mean +/- standard deviation, and categorical variables as headcounts and percentages. Statistical analyses will be performed using jamovi 2.3.18 software with a threshold α = 0.05.

Quantitative analysis

After checking for applicability, in order to evaluate the effectiveness of the intervention in the experimental group compared to the control group, a MANOVA will be performed. The dependent variables are anxiodepressive symtoms, pain, quality of life and fatigue, and the independent variables are the different measurement times. The investigators will control for age, gender, socioeconomic status, diagnosis absorption, dissociation, and amusement, . If suitable, the investigators will make post-hoc comparisons to compare scores between groups and at each measurement time with a Bonferroni correction.

Correlations will be performed on variables measured during the transplant phase (anxiety, pain, fatigue, absorption, dissociation, amusement) to measure the immediate effects of VRH. Correlations will be made between pre- and post-intervention scores and will be estimated with Pearson's or Spearman's correlation and their 95 % CI. Correlations will also be made between primary and secondary outcomes.

The investigators expect better effects on primary outcomes, i.e., diminution of anxiety and pain levels and secondary outcomes, i.e., quality of life and fatigue for the VRH program than for condition C.

Qualitative analysis

The verbatims from the semi-structured interviews will be analyzed qualitatively using NVivo software. The software enables thematic content analysis, highlighting codes in the text and graphically grouping them into themes to create a thematic tree. To identify the key themes in patients' explicit discourse, a general inductive method inspired by Braun and Clarke (2021) will be employed, aiming to uncover recurring patterns directly from the data. This data-driven approach involves deriving themes organically from the dataset. The recommended process involves six main steps after preparing the raw data files (e.g., formatting and correcting transcription errors): 1) thoroughly reading the transcripts to become familiar with the data, 2) conducting line-by-line coding to generate initial codes, 3) identifying recurring themes, 4) reviewing and refining these themes, 5) defining and naming each theme, and 6) producing a report that incorporates verbatim examples.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Suffering from multiple myeloma or lymphoma eligible for transplant
* Understanding French

Exclusion Criteria:

* Deafness
* Blindness
* Confusion or psychopathological disorders (for example, schizophrenia) that may impair communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Anxiety and depression | Studied one week, one month and three months post-transplantation
  Anxiety-depression will be measured using the Hospital anxiety and depression scale (HADS), a scale validated in French for cancer. This scale is made up of 14 items: 7 items determine the degree of anxiety and the other 7, the degree of depression. The score of each subscale is calculated by summing the score of each item, which varies between 0 and 3, so that each subscale can reach a maximum score of 21
Level of pain | Studied one week, one month and three months post-transplantation
  Pain will be assessed with the Brief Pain Inventory. This scale is made of 8 items on a 10-points Lickert scale (0=no pain, 10=worst pain) assessing severity of pain, impact of pain on daily function, location of pain, pain medications and amount of pain relief in the past 24 hours or the past week.

SECONDARY OUTCOMES:
Level of quality of life | Studied one week, one month and three months post-transplantation
  Quality of life will be assessed by FACT-BMT, which comprises 50 items in 5 subscales : Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, Bone Marrow Transplantation Subscale scored on a 5-points Likert scale (0=not at all, 4=very much).
Absorption | Studied immediately before and after each use of the intervention 4 times during the two weeks in possession of the VR headset.
  Absorption will be measured using a eleven-level Visual Numerical Scales (VNS) (minimum 0=no absoption at all, maximum 10=totally absorbed)
Dissociation | Studied immediately before and after each use of the intervention 4 times during the two weeks in possession of the VR headset.
  Dissociation will be measured using a eleven-level Visual Numerical Scales (VNS) (minimum 0=no dissociation, maximum 10=fully dissociated).
Level of expectation and satisfaction | Measured respectively one week post-transplantation and three months post-transplantation
  Level of expectation and satisfaction will be assessed using a five-level Visual Numerical Scales (VNS) (1 = "not at all satisfied", 5 = "very satisfied") and semi-structured interviews
Cybersickness | Measured after each use of the intervention 4 times during the two weeks in possession of the VR headset.
  Cybersickness will be measured using the Simulator Sickness Questionnaire (SSQ), a scale validated in French assesses cybersickness symptoms related to VR immersion. It contains 16 items divided in two subsacles: nausea and oculomotor, which the participant must qualify with "not at all" (scored 0) , "a little" (scored 1), "moderately" (scored 2) or "severely" (scored 3).
Amusement | Studied immediately before and after each use of the intervention 4 times during the two weeks in possession of the VR headset.
  Amusement will be measured using a eleven-points Visual Numerical Scales (VNS) (minimum 0=no amusement, maximum 10=very amused)
Level of pain | Studied immediately before and after each use of the intervention 4 times during the two weeks in possession of the VR headset.
  Pain will be assessed using a Visual Numerical Scales (VNS) (minimum 0=no pain at all, maximum 10=very painful)
Fatigue | Studied one week, one month and three months post-transplantation
  Fatigue will be assessed with the Multidimensional Fatique Inventory 10 items version (MFI-10), a scale adapted for cancer. It is scored on a 5-points Likert Scale going form minimum 1: "do not agree at all" to maximum 5: "totally agree".
Anxiety | Studied immediately before and after each use of the intervention 4 times during the two weeks in possession of the VR headset.
  Anxiety will be measured using a eleven-level Visual Numerical Scales (VNS) (minimum 0=not anxious at all, maximum10= very anxious)
Fatigue | Studied immediately before and after each use of the intervention 4 times during the two weeks in possession of the VR headset.
  Fatigue will be measured using a ten-level Visual Numerical Scales (VNS) (minimum 0= no fatigue at all, maximum 10=very fatigued)
Relaxation | Studied immediately before and after each use of the intervention 4 times during the two weeks in possession of the VR headset.
  Relaxation will be measured using a eleven-points Visual Numerical Scales (VNS) (minimum 0=not relaxed at all, maximum 10=relaxed)

CONTACTS AND LOCATIONS:
Overall Officials: David Ogez, Ph.D, Principal Investigator — Université de Montréal
Locations (1):
- Centre de Recherche de l'Hôpital Maissonneuve-Rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared in a dedicated OSF repository.
Supporting Information: Study Protocol, SAP
Time Frame: Supporting information will be available from the definitive publication of results.
Access Criteria: All IPD that underlie results in a publication will be shared in a dedicated OSF repository,